CLINICAL TRIAL: NCT05066308
Title: Evaluation of Cannabidiol for Reduction of Brain Neuroinflammation
Brief Title: Cannabidiol for Reduction of Brain Neuroinflammation
Acronym: CBD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jodi Gilman, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2021P002617
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Back Pain; Depressive Symptoms
Keywords: back pain; depression; depressive symptoms; cannabis; cannabidiol
MeSH Terms: conditions — Back Pain; Depression; Marijuana Abuse | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (CBD) (Experimental): The recommended starting dosage is 2.5mg/kg taken twice daily. The titration schedule recommended in the EPIDIOLEX label will be followed, with 2.5 mg/kg twice daily in week 1, 5 mg/kg twice daily in week 2, 7.5 mg/kg twice daily in week 3, and 10 mg/kg twice daily in week 4 with the second PET scan conducted after one week at the maximum labeled dose. Any participant not tolerating a given dose can either go back down to the next lowest dose or delay uptitration at any week in the protocol. Participants will be instructed to take Epidiolex with a meal rather than in a fasted state. Participants will be treated for 4 weeks in total.
  Interventions: Drug: CBD
- Placebo (Placebo Comparator): The placebo will be taken at identical doses to the active drug condition.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CBD — Epidiolex, an agent within the anti-epileptic drug class, will be used. Epidiolex, Greenwich Biosciences Inc.'s CBD formulation, is a 100 mg/mL purified oral solution, dissolved in the excipients sesame oil and anhydrous ethanol with added sweetener (sucralose) and strawberry flavoring. The drug is formulated from extracts prepared from Cannabis sativa L. plants that have a defined chemical profile and contain consistent levels of CBD as the principal phytocannabinoid. Extracts from these plants are processed to yield pure (>95%) CBD that typically contains less than 0.5% (w/w) THC. Cannabidiol is the active ingredient in Epidiolex; inactive ingredients include dehydrated alcohol, sesame seed oil, strawberry flavor, and sucralose. Of note, CBD has no psychoactive properties.
  Other Names: Epidiolex
  Arms: Cannabidiol (CBD)
Other: Placebo — Placebo CBD will be identical to the active CBD, a 100 mg/mL purified oral solution, dissolved in the excipients sesame oil and anhydrous ethanol with added sweetener (sucralose) and strawberry flavoring, but with no CBD.
  Arms: Placebo

SUMMARY:
This study will investigate whether cannabidiol (CBD), the primary centrally and peripherally active non-intoxicating compound in the cannabis plant, exerts anti-neuroinflammatory effects in patients with chronic low back pain (cLBP) with or without mild-to-moderate depression.

DETAILED DESCRIPTION:
This is a randomized, double-blind, 2-arm mechanistic trial that seeks to assess the effects of CBD and placebo in patients with cLBP with and without mild-to-moderate depression, using integrated positron emission tomography / magnetic resonance imaging (PET/MRI) scans. The use of integrated PET/MRI will make it possible to simultaneously evaluate neuroinflammation (using [11C]PBR28, a second-generation radioligand for TSPO) and striatal function (using the Monetary Incentive Delay task, a validated fMRI task that probes behavioral and neural responses to rewards and losses).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75;
2. The ability to give written, informed consent;
3. Fluency in English;
4. Average worst daily pain of at least 4 on a 0-10 scale of pain intensity, during a typical day. Pain needs to be present for at least 50% of days during a typical week;
5. On a stable pain treatment (pharmacological or otherwise) for the previous four weeks;
6. Diagnosis of chronic low back pain, ongoing for at least 6 months prior to enrollment.
7. High or mixed affinity binding to [11C]PBR28 identified by the Ala147Thr TSPO polymorphism in the TSPO gene (rs6971)

Exclusion Criteria:

1. Outpatient surgery within 2 weeks and inpatient surgery within 1 month of the time of scanning (this timeframe may be extended if they are not fully recovered from the surgery);
2. Elevated baseline transaminase (ALT and AST) levels above 3 times the Upper Limit of Normal (ULN), accompanied by elevations in bilirubin above 2 times the ULN;
3. Any interventional pain procedures within 6 weeks prior to scanning procedure or at any point during study enrollment;
4. Surgical intervention or introduction/change in opioid regimen at any point during study enrollment;
5. Contraindications to fMRI scanning and PET scanning (including presence of a cardiac pacemaker or pacemaker wires, metallic particles in the body, vascular clips in the head or previous neurosurgery, prosthetic heart valves, claustrophobia);
6. Implanted spinal cord stimulator (SCS) for pain treatment;
7. Any history of neurological illness or major medical illness, unless clearly resolved without long-term consequences;
8. Current or past history of major psychiatric illness (PTSD, depression, and anxiety are exclusion criteria only if the conditions were so severe as to require hospitalization in the past year);
9. Harmful alcohol drinking as indicated by an AUDIT score ≥ 16;
10. Pregnancy or breast feeding;
11. History of head trauma requiring hospitalization;
12. Major cardiac event within the past 10 years;
13. Regular use of recreational drugs in the past 3 months;
14. Use of cannabis-containing products, such as products containing THC or over the-counter or dispensary CBD, for 2 weeks prior to starting the study medication and during the 4 weeks of taking the study medication;
15. Use of immunosuppressive medications, such as prednisone, TNF medications within 2 weeks of the visit;
16. Current bacterial or viral infection likely affecting the central nervous system;
17. Epilepsy;
18. Use of the medications valproate and clobazam, which may increase risk of hepatic AEs;
19. Safety concerns related to use of any of the following medications will be discussed on an individualized basis with a physician:

    * Strong and moderate CYP3A4 inhibitors including boceprevir, cobicistat, conivaptan, danoprevir, elvitegravir, ritonavir, indinavir, itraconazole, ketoconazole, lopinavir, paritaprevir and ombitasvir and/or dasabuvir, posaconazole, saquinavir and telaprevir, tipranavir, clarithromycin, diltiazem, idelalisib, nefazodone, nelfinavir, troleandomycin, voriconazole, aprepitant, cimetidine, ciprofloxacin, clotrimazole, crizotinib, cyclosporine, dronedarone, erythromycin, fluconazole, fluvoxamine, imatinib, tofisopam, disulfiram, and verapamil;
    * Strong and moderate inhibitors of CYP2C19 including fluoxetine and ticlopidine;
    * Sensitive and moderately sensitive substrates of CYP2C19 including clobazam, lansoprazole, omeprazole, S-mephenytoin, and rabeprazole;
    * Sensitive and moderately sensitive substrates of CYP1A2 including alosetron, duloxetine, ramelteon, tasimelteon, theophylline, tizanidine, pirfenidone, and ramosetron;
    * Sensitive and moderately sensitive substrates of CYP2B6 including bupropion and efavirenz;
    * Sensitive and moderately sensitive substrates of CYP2C8 including repaglinide, montelukast, pioglitazone, and rosiglitazone;
    * Sensitive and moderately sensitive substrates of CYP2C9 including tolbutamide, celecoxib, glimepiride, and warfarin;
    * Sensitive and moderately sensitive substrates of UGT1A9 including diflunisal, propofol, and fenofibrate;
    * Sensitive and moderately sensitive substrates of UGT2B7 including, gemfibrozil, lamotrigine, and morphine;
20. CNS depressants including all antipsychotics, benzodiazepines (except for alprazolam, clonazepam, and lorazepam, which have low binding affinity to TSPO44-48), and non-benzodiazepine sleep aids that have a known unsafe reaction with CBD;
21. Use of opioids ≥ 30 mg morphine equivalents on average per month;
22. Actively suicidal, history of suicide attempt or an aborted attempt within the last 5 years, or engagement in non-suicidal self-injurious behavior within the last year;
23. Allergy to sesame oil, and any other ingredients of EPIDIOLEX;
24. Any other contraindications to CBD administration noted by the study physician;
25. Any significant change in drug use and pain treatment from screening visit;
26. In the opinion of the investigators, unable to safely participate in this study and/or provide reliable data (e.g., unable to reliably rate pain; unlikely to remain still during the imaging procedures, etc).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Changes in Neuroinflammation in the Thalamus | Change from Baseline to Week 4
  The investigators will test for the presence of a significant treatment effect in the brain [11C]PBR28 signal in the thalamus, in order to test whether patients in the CBD arm will demonstrate significantly larger treatment-related reductions in neuroinflammation, compared to patients in the placebo arm.

SECONDARY OUTCOMES:
Changes in Neuroinflammation in Limbic Regions | Change from Baseline to Week 4
  The investigators will test for the presence of a significant treatment effect in the brain [11C]PBR28 in limbic regions (pgACC, aMCC), in order to test whether patients in the CBD arm will demonstrate significantly larger treatment-related reductions in neuroinflammation, compared to patients in the placebo arm.
Correlation Between Reductions in Thalamic [11C]PBR28 PET Signal and Reductions in Clinical Pain Ratings | Change from Baseline to Week 4
  The investigators will test whether reductions in thalamic [11C]PBR28 PET signal correlate with reductions in clinical pain ratings, as assessed by the "worst pain" item of the Brief Pain Inventory - Short Form. The "worst pain" item's scale ranges from 0 - 10, with a higher score indicating worse pain intensity.
Correlation Between Reductions in Limbic [11C]PBR28 PET Signal and Reductions in Depressive Symptoms | Change from Baseline to Week 4
  The investigators will test whether reductions in pgACC/aMCC [11C]PBR28 PET signal (as measured by Standardized Uptake Value Ratio) correlate with reductions in depressive symptoms, as measured by the Beck Depression Inventory-II. The Beck Depression Inventory-II scale ranges from 0 - 63, with a higher score indicating greater depression.
Change in Clinical Pain Ratings | Change from average score during the 7 days prior to treatment (Baseline) to average score during the final week of treatment
  The "worst pain" item of the Brief Pain Inventory - Short Form will be used daily to assess pain intensity. The scale ranges from 0 - 10, with a higher score indicating worse pain intensity.
Change in Pain Bothersomeness | Change from average score during the 7 days prior to treatment (Baseline) to average score during the final week of treatment
  Pain bothersomeness will be assessed daily on a scale from 0 - 10, with a higher score indicating greater bothersomeness.
Change in Depressive Symptoms | Change from Baseline to Week 4
  The Beck Depression Inventory-II will be used to assess symptoms of depression. The scale ranges from 0 - 63, with a higher score indicating greater depression.
Patient Global Impression of Change | Week 4
  The Patient Global Impression of Change scale will be used to assess participants' perceptions about their global improvement related to their low back pain. The scale ranges from 0 - 7, with a higher score indicating greater overall improvement.

OTHER OUTCOMES:
Change in Functional Brain Reward Circuitry [Exploratory] | Change from Baseline to Week 4
  The Monetary Incentive Delay task will be used to assess striatal response to the anticipation and/or consumption of rewards/losses.
Change in Pain Severity & Interference with Daily Functioning [Exploratory] | Change from Baseline to Week 4
  The full Brief Pain Inventory - Short Form will be used to assess pain severity and its interference with daily functioning. Pain severity is assessed on a scale from 0 - 10, with a higher score indicating more severe pain. Daily functioning is also assessed on a scale from 0 - 10, with a higher score indicating that pain more greatly interferes with functioning.
Change in Pain Catastrophizing [Exploratory] | Change from Baseline to Week 4
  The Pain Catastrophizing Scale will be used to assess pain catastrophizing. The scale ranges from 0 - 52, with a higher score indicating greater catastrophic thinking.
Change in Neuropathic Pain Components [Exploratory] | Change from Baseline to Week 4
  The PainDETECT questionnaire will be used to assess neuropathic components of pain. The scale ranges from -1 to 38, with a higher score indicating more neuropathic-like symptoms.
Change in Disability Related to Low Back Pain [Exploratory] | Change from Baseline to Week 4
  The Oswestry Disability Index will be used to assess disability related to low back pain. The scale ranges from 0 - 50, with a higher score indicating greater disability.
Change in Widespread Pain and Fibromyalgia Symptom Severity [Exploratory] | Change from Baseline to Week 4
  The American College of Rheumatology's fibromyalgia survey will be used to assess widespread pain and fibromyalgia symptom severity. The widespread pain subscale ranges from 0 - 19, with a higher score indicating more widespread pain. The fibromyalgia symptom severity subscale ranges from 0 - 12, with a higher score indicating more severe symptoms.
Change in Depression [Exploratory] | Change from average score of the 7 days prior to initiation of treatment to average score of the 7 days of Week 4
  In addition to the secondary outcome which uses the BDI-II to assess change in depression, depression will also be assessed daily on a scale from 0 - 10, with a higher score indicating greater depression.
Change in Health-Related Quality of Life [Exploratory] | Change from Baseline to Week 4
  The Patient-Reported Outcomes Measurement Information System(PROMIS)-29 will be used to assess health-related quality of life, including physical, mental, and social health. The scale uses a t-score metric. For positively worded measures, a higher t-score indicates greater health within that domain; for negatively worded measures, a higher t-score indicates poorer health within that domain.
Change in Sleep Quality [Exploratory] | Change from Baseline to Week 4
  The Pittsburgh Sleep Quality Index will be used to assess sleep quality. The scale ranges from 0 - 21, with a higher score indicating less healthy sleep quality.
Change in Widespreadness of Pain Sensation [Exploratory] | Change from Baseline to Week 4
  The SymptomMapper app, a digital tablet-based application where patients can mark where on the body they are experiencing pain, will be used to assess widespreadness of pain sensation.
Change in Spinal Cord TSPO Signal [Exploratory] | Change from Baseline to Week 4
  The investigators will test whether reductions in spinal cord [11C]PBR28 PET signal correlate with reductions in clinical pain ratings, as assessed by the "worst pain" item of the Brief Pain Inventory - Short Form. The "worst pain" item's scale ranges from 0 - 10, with a higher score indicating worse pain intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All data, code, and materials used in the analyses can be provided by Jodi Gilman and Marco Loggia and Massachusetts General Hospital pending scientific review and a completed data use agreement/material transfer agreement beginning one year after publication of the results. Requests for all materials should be submitted to Jodi Gilman at jgilman1@mgh.harvard.edu or to Marco Loggia at marco.loggia@mgh.harvard.edu.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available beginning one year after publication of the results.
Access Criteria: Data will be provided pending a scientific review and a completed data use agreement/material transfer agreement. Requests should be submitted to Jodi Gilman at jgilman1@mgh.harvard.edu or to Marco Loggia at marco.loggia@mgh.harvard.edu

REFERENCES:
- [Derived] Pike CK, Kim M, Schnitzer K, Mercaldo N, Edwards R, Napadow V, Zhang Y, Morrissey EJ, Alshelh Z, Evins AE, Loggia ML, Gilman JM. Study protocol for a phase II, double-blind, randomised controlled trial of cannabidiol (CBD) compared with placebo for reduction of brain neuroinflammation in adults with chronic low back pain. BMJ Open. 2022 Sep 19;12(9):e063613. doi: 10.1136/bmjopen-2022-063613. PMID 36123113

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/08/NCT05066308/SAP_000.pdf